CLINICAL TRIAL: NCT02071966
Title: Effects of TIcaGREloR on Circulating Microparticles and Micro-RNAs in Patients With Non ST Elevation Acute Coronary Syndromes
Brief Title: Study of Effects of Ticagrelor on Microparticles and Micro-RNA in NSTE-ACS
Acronym: TIGER-M
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: slow enrollment
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, L.M. Biasucci, Professor, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D5130L00028
Record Dates: First submitted 2014-02-21; First posted 2014-02-26 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Non ST Segment Elevation Acute Coronary Syndrome
Keywords: Micro-RNA, Microparticles, Ticagrelor, NSTE-ACS
MeSH Terms: interventions — Ticagrelor; Clopidogrel

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ticagrelor (Active Comparator): Ticagrelor: oral, 180 mg once for the first dose then 90 mg twice a day
  Interventions: Drug: Ticagrelor
- Clopidogrel (Active Comparator): Clopidogrel: oral, 300 or 600 mg once for the first dose, 75 mg once a day
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Ticagrelor — Comparison of Ticagrelor with another anti-platelet drug (Clopidogrel)
  Other Names: Brilique
  Arms: Ticagrelor
Drug: Clopidogrel — Comparison of Clopidogrel with another anti-platelet drug (Ticagrelor)
  Other Names: Plavix
  Arms: Clopidogrel

SUMMARY:
The aim of the study is to learn more about the pathophysiology of acute coronary syndrome (ACS) and to evaluate the mechanisms responsible of the action and benefits of ticagrelor.

Ticagrelor is an oral and reversible inhibitor of P2Y12 receptor. Few information is available about the action of ticagrelor on the molecules involved in thrombogenesis and platelets activation in ACS.

The aim of this study is to evaluate the mechanisms of ticagrelor action in vivo.

It was observed that patients with myocardial infarction have higher blood levels of microparticles than patients with unstable angina or stable angina.

The investigators assumed that ticagrelor benefits are represented by a reduction of microparticle levels, a marker of endothelial dysfunction in patients with cardiovascular disease, and by a modification in microRNAs pattern, fragments of mRNA that have a regulatory action in various cellular processes (such as proliferation, differentiation, growth and cellular death) and represent new biomarkers in ACS.

DETAILED DESCRIPTION:
Ticagrelor is an oral, reversibly binding P2Y12 receptor inhibitor that yields, in a dose-dependent fashion, greater and more consistent inhibition of platelet aggregation than standard regimens of clopidogrel in patients with stable atherosclerotic disease and ACS. However, little information is available regarding its complex effect on thrombogenesis and platelet activation in acute coronary syndromes setting. It has been widely demonstrated the potential role of MP in several biologic processes known to take part to pathophysiology of coronary syndromes, such as inflammation, coagulation and apoptosis. Recent studies focused on miRNAs' regulatory activity of several cellular processes, such as proliferation, differentiation, development, and cell death, and on their role as biomarkers in ACS. The investigators suppose that the observed major efficacy of ticagrelor is related to its actions on MP and microRNAs. Considering the major clinical effectiveness shown by ticagrelor in comparison with clopidogrel, the investigators hypothesize a more pronounced MP levels reduction as a possible mechanism for ticagrelor clinical benefits. Moreover, on the basis of the last evidences of microRNA involvement in the ACS pathophysiology, the investigators aim to assess the effect of ticagrelor on microRNA expression, in order to provide evidences for pleiotropic actions of this drug, which could partially explain its major efficacy in reduction of cardiovascular events in ACS patients.

In summary, principal hypothesis of the study are:

* Considering that ticagrelor is a stronger P2Y12 receptor inhibitor than clopidogrel, the investigators suppose that an increased inhibition of P2Y12 receptor by ticagrelor could reduce circulating levels of platelet and endothelial MP.
* In consideration of the observed role of microRNAs in expression of P2Y12 receptor, the investigators speculate that patient's susceptibility to P2Y12 receptor inhibitors could be influenced by microRNAs levels. Moreover, the investigators suppose that ticagrelor could influence microRNAs levels, considered as marker of cardiovascular risk

Aims of the study are:

* to assess MP levels variation in Non ST-Elevation Acute Coronary Syndromes (NSTE-ACS) patients treated with ticagrelor in addition to low or high acetyl-salicylic acid (ASA), in comparison with clopidogrel+ASA treatment, to demonstrate that major clinical efficacy of ticagrelor could be partially attributed to its influence on release of MP, that have an important role in coronary instability.
* to evaluate microRNAs levels variation in Non ST-Elevation Acute Coronary Syndromes (NSTE-ACS) patients treated with ticagrelor in addition to low or high ASA, in comparison with clopidogrel+ASA treatment, and to study possible correlations between microRNAs and MP levels, supposing that the ability of ticagrelor in reduced MP level could be related with microRNAs expression.

ELIGIBILITY:
Inclusion Criteria:

* NSTE-ACS
* Male, 50-80 years old
* Female, postmenopausal age

Exclusion Criteria:

* Female, premenopausal age
* autoimmune disease
* infectious disease
* neoplasms
* diabetes
* chronic renal failure
* moderate or severe liver insufficiency
* GRACE risk score>140
* ACS or cerebrovascular accidents in previous three months
* in-stent restenosis
* surgery or trauma in previous three months
* active bleeding
* fibrinolytic therapy within 24 hours before randomization
* need for oral anticoagulation therapy
* an increased risk of bradycardia
* drugs study hypersensitivity (including aspirin)
* co-administration of ticagrelor or clopidogrel with strong CYP3A4 inhibitors

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2012-11; Primary Completion 2015-12 (Actual); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Micro-RNA and microparticles | up to three months

CONTACTS AND LOCATIONS:
Overall Officials: Luigi M Biasucci, Professor, Principal Investigator — Catholic University of the Sacred Heart
Locations (1):
- Policlinico "A.Gemelli", Rome, Italy